CLINICAL TRIAL: NCT01295450
Title: A Clinical Multicenter, Phase III, Randomized, Double-blind, Prospectively to Evaluate the Efficacy and Tolerability of Apevinat BC Compared to Vitamin Complex in Stimulating the Appetite
Brief Title: Study to Evaluate the Efficacy and Tolerability of Apevinat BC Compared to Vitamin Complex
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MDCPharma Produtos Farmaceuticos LTDA (Industry)
Responsible Party: MDCPharma Produtos Farmaceuticos LTDA, Industry
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDC-APEVINAT-01/10
Record Dates: First submitted 2011-01-19; First posted 2011-02-14 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Lack of Appetite; Anorexia
Keywords: Phase III; Apevinat BC; Lack of appetite
MeSH Terms: conditions — Anorexia | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin Complex (Active Comparator): A vitamin complex contains: B1, B2, B3, B3 and C vitamins. Administer the recommended dosage preferably one hour before meals: 5 ml three times daily.
  Interventions: Drug: Apevinat BC
- Apevinat BC (Experimental): Apevinat BC presents in its formula the cyproheptadine hydrochloride (0,800 mg), tiamin hydrochloride(0,120 mg), Riboflavin sodium phosphate (0,200 mg), nicotinamide (1,334 mg, piridoxin hydrochloride (0,134 mg), ascorbic acid (4,334 mg).
  Administer the recommended dosage for children 7 to 14, preferably one hour before meals: 5 ml three times daily.
  Interventions: Drug: Vitamin Complex

INTERVENTIONS:
Drug: Apevinat BC — Apevinat BC presents in its formula the cyproheptadine hydrochloride (0,800 mg), tiamin hydrochloride(0,120 mg), Riboflavin sodium phosphate (0,200 mg), nicotinamide (1,334 mg, piridoxin hydrochloride (0,134 mg), ascorbic acid (4,334 mg).
  Administer the recommended dosage for children 7 to 14, preferably one hour before meals: 5 ml three times daily.
  Other Names: MDCPharma
  Arms: Vitamin Complex
Drug: Vitamin Complex — A vitamin complex contains: B1, B2, B3, B3 and C vitamins. Administer the recommended dosage preferably one hour before meals: 5 ml three times daily.
  Other Names: Polivitamin, B and C Complex.
  Arms: Apevinat BC

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of Apevinat BC compared to vitamin complex, in the treatment of lack of appetite and prevention of deficiency of B and C vitamins.

DETAILED DESCRIPTION:
Apevinat BC presents in its formula the cyproheptadine hydrochloride, which is an antihistamine and anti-serotonin with stimulant of appetite property associated with the vitamin B complex and C, in balanced amounts.

This combination is specially formulated to adequately serve patients with anorexia represented by lack of appetite or appetite diverted to diets without the necessary vitamins. For the anorexic patients that are common B and C hypovitaminosis, the use of Apevinat BC will have a synergistic and joint action to increase appetite and facilitate correction of a diet while also supplement with B and C vitamins, this association does not decreases its tolerability and safety but hits adequately the purpose of therapeutic orexigenic.

The current study will compare the efficacy and tolerability of Apevinat BC to vitamin complex administered three times a day, in the prevention and treatment of lack of appetite and B and C hypovitaminosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presents lack of appetite;
* Wash out 20 days after ingestion before similar drug;
* Responsible for the least able to understand and maintain their adherence to protocol;
* Patients of all ethnic groups of both sexes, aged 7-14 years;
* Responsible for the minor must consent to participate in the same study, through the signing of consentiment term;
* Responsible for the minor should be able to understand the proper use of medication;

Exclusion Criteria:

* Patients with parasitic infections;
* Patients with angle closure glaucoma or open;
* Patients with a predisposition to urinary retention;
* Patients with peptic ulcer or stenotic pylorus-duodenal obstruction;
* debilitated patients or in acute asthma attack;
* Patients who have poor appetite caused by any serious illness;
* Patients who are taking any medications that depress the central nervous system;
* Patients who take medication monoamine oxidase inhibitors, tricyclic antidepressants, phenothiazine, probenecid, levodopa, phenytoin, phenobarbital, chloramphenicol, cyclophosphamide, cyclosporine, chlorambucil, corticotrophin, mercaptopurine, isoniazid, penicillin, estrogens, contraceptives, haloperidol, ipatrópico, barbiturates, Primidone, salicylates;
* Patients with known hypersensitivity to any components of the formula;
* Patients who are participating in another clinical trial;
* Inability to compliance with the protocol;
* Any condition that in the opinion of the investigator would prohibit the inclusion and patient compliance with the protocol.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of Apevinat BC in appetite stimulation. | 30 days
  Evaluate the efficacy of BC Apevinat in appetite stimulation compared to vitamins.

SECONDARY OUTCOMES:
Evaluate the tolerability of Apevinat BC in appetite stimulation. | 30 days
  To evaluate the tolerability of Apevinat BC in appetite stimulation compared to vitamins.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim CS D' Azevedo, Investigator, Principal Investigator — A/Z Clinical; Felicio S Neto, Investigator, Principal Investigator — Dr. Felicio Savioli Clinical
Locations (1):
- ABC School of Medicine, São Paulo, São Paulo, Brazil